CLINICAL TRIAL: NCT02767583
Title: Assessment of the Prevalence of Small Fiber Peripheral Neuropathy Among Non-diabetic Obese Patients
Acronym: NEUROBISITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Neuropathies and obesity
Record Dates: First submitted 2016-05-04; First posted 2016-05-10 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Neuropathology
Keywords: Neuropathology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non diabetic obese (Experimental): Non diabetic obese with BMI 35-55 kg / m2 consulting for the first time at the Centre of obesity of Paris Saint Joseph Hospital Group will got a themotest and Sudoscan exams de determine their neuropathology.
  Interventions: Device: Exams

INTERVENTIONS:
Device: Exams — Patients the eligibility criteria will be proposed at the first consultation in central obesity, participate in a clinical study to assess the prevalence of subclinical damage peripheral nerves by simple and painless rapid measurement of skin conductance on the palm of the feet with the Sudoscan® device during the consultation and a Thermotest®, as well as monitoring during the various follow-up consultation after any bariatric surgery or not. This monitoring will be done by the same neurophysiological tests.

SUMMARY:
Background / rational:

Obesity is associated with significant comorbidities including type 2 diabetes (insulin resistance), heart disease, stroke, hypertension, sleep apnea syndrome, dyslipidemia, cancer, hepatobiliary diseases, orthopedic complications and psychosocial impact 1 .

Peripheral neuropathy is a known complication in the type I and II diabetes and glucose intolerance and metabolic syndrome in 2. Outside of diabetes (type I and II) that are associated with cardiovascular risk high vascular, presence of metabolic syndrome constitutes in itself a well demonstrated vascular risk factor. Its definition requires the presence of three elements from the following 5: abdominal obesity (high waist circumference), high blood pressure, high fasting blood sugar, high triglycerides and / low HDL-cholesterol 3.

This peripheral neuropathy predominantly affects sensory fibers of small poorly myelinated diameter (Aδ fibers and C) and autonomous sensory fibers and is called small fiber neuropathy 4. The cardinal sign of NAION is the presence of neuropathic pain but abnormalities in physical examination are often absent and conventional electromyography is faulted to make the diagnosis. These small fibers are also constituent of the autonomic nervous system and causes damage autonomic dysfunction that can manifest the cardiovascular system (hypotension, cardiac conduction disorders), digestive, sweat, sphincter. neuropathy of the diagnosis of small fibers is suggested clinically by the presence of neuropathic pain often contrasting with a normal clinical examination. The confirmation is based on electrophysiology with various techniques and quantification of intra-epidermal nerve fibers.

Main objective / secondary:

Primary objective :

To determine the prevalence of a small fiber peripheral neuropathy in nondiabetic obese patients, by measuring skin conductance ion Chlorine (Sudoscan®) evaluating small fibers C autonomic

Secondary objectives:

* Evaluation of the prevalence of occurrence of peripheral neuropathy by Sudoscan® during follow-up after treatment of obese patients with bariatric surgery (months) M1, 3, 6, 9, 12.
* Correlation of results obtained Sudoscan® quantitative sensory testing (QST) Thermotest® evaluating small sensory fibers Aδ, among non-operated non-diabetic obese patients and in the postoperative follow-up (months) M1, 3, 6, 9, 12.
* Characterization of electromyographic parameters (motor and sensory conduction) in patients with a skin conductance measured by lowered Sudoscan® and / or a threshold of sensitivity to pain increased Thermotest®.
* Correlation between the presence of a small fiber neuropathy in non-diabetic obese subjects with clinical and biological parameters collected.

Methodology Design: prospective, single-center Study duration: 24 months (estimate: 3-5 patients included / week of 15 patients collected in central obesity / week) including 12 months of inclusion.

Number of topics to include: 100 over a period of one year to adjust to the rhythm of the inclusions.

As mentioned, patients will be a measure of impedance of the skin to products chlorine ions by the sweat glands via the Sudoscan®, marketed and used among diabetic patients or not for the detection of violations neuropathic (cf. references and CE certificate attached to the dossier).

The Thermotest® is also marketed and used in diabetic and non-diabetic patients (see references and CE certificate attached to the dossier).

Our center has gained experience of these techniques for the detection of peripheral neuropathy in several patient populations (diabetes and cancer in particular); manipulators (doctors and technicians) are trained in these techniques.

DETAILED DESCRIPTION:
Main objective / secondary:

Primary objective :

To determine the prevalence of a small fiber peripheral neuropathy in nondiabetic obese patients, by measuring skin conductance ion Chlorine (Sudoscan®) evaluating small fibers C autonomic

Secondary objectives:

* Evaluation of the prevalence of occurrence of peripheral neuropathy by Sudoscan® during follow-up after treatment of obese patients with bariatric surgery (months) M1, 3, 6, 9, 12.
* Correlation of results obtained Sudoscan® quantitative sensory testing (QST) Thermotest® evaluating small sensory fibers Aδ, among non-operated non-diabetic obese patients and in the postoperative follow-up (months) M1, 3, 6, 9, 12.
* Characterization of electromyographic parameters (motor and sensory conduction) in patients with a skin conductance measured by lowered Sudoscan® and / or a threshold of sensitivity to pain increased Thermotest®.
* Correlation between the presence of a small fiber neuropathy in non-diabetic obese subjects with clinical and biological parameters collected.

Inclusion / non-inclusion:

Inclusion criteria:

morbidly obese patients:

* BMI 35-55 kg / m²,
* Male or female,
* Age> 18 and <60 years,
* Consultant for the first time at the Centre of obesity of Paris Saint Joseph Hospital Group.

Exclusion criteria:

* Diabetes known treaty
* Co-morbidity related to obesity: heart disease, respiratory failure
* Other causes of peripheral neuropathy:

  * Alcohol Poisoning
  * Renal failure (clearance ≤ 60 mL / min)
  * Infection HIV, hepatitis B, C
  * Deficiencies vitamins B1, B6, B12, folate
  * Treatment with vitamin B6
  * thyroid disease antecedent
  * Previous history of autoimmune disease
  * Previous history of cancer
  * Previous history of neurotoxic treatment (chemotherapy, etc. see list provided in annex)
  * ICU hospitalization antecedent> 48 hours.
  * known history of peripheral neuropathy.

Development of the study:

If patients the eligibility criteria, it will be proposed at the first consultation in central obesity, participate in a clinical study to assess the prevalence of subclinical damage peripheral nerves by simple and painless rapid measurement of skin conductance on the palm of the feet with the Sudoscan® device during the consultation and a Thermotest®, as well as monitoring during the various follow-up consultation after any bariatric surgery or not. This monitoring will be done by the same neurophysiological tests.

* During the preoperative assessment that will be conducted in the planned hospital in Diabetology Service, written information will be given to patient and no objection will be drawn, then the following tests will be done:
* The measurement of skin conductance by Sudoscan® and the extent of the painful sensitivity to temperature Thermotest® will be made for all patients included in the study.
* If the records Sudoscan® skin conductance less than 60μS, we propose a Electroneuromyography the patient as usual on GHPSJ.
* Measurement of weight, height, waist circumference and hip circumference patient
* The DN4 scale and Uens clinical neuropathy score.
* A measurement of blood pressure will be
* A biological sample will be taken on an empty stomach.
* For patients with plantar skin conductance will be lowered <60μSiemens and / or whose pain threshold will warm significantly elevated (Thermotest®), if necessary electromyogram will be realized in the second time (appointment given to the output consultation with the endocrinologist.
* During the postoperative follow-up usually expected for this type of surgery, 1, 3, 6, 9 and 12 months will be made the same clinical examinations than those made during the preoperative assessment and the type of surgery performed. Laboratory tests will be carried out in the usual care for surgical patients.

Methodology Design: prospective, single-center Study duration: 24 months (estimate: 3-5 patients included / week of 15 patients collected in central obesity / week) including 12 months of inclusion.

Number of topics to include: 100 over a period of one year to adjust to the rhythm of the inclusions.

As mentioned, patients will be a measure of impedance of the skin to products chlorine ions by the sweat glands via the Sudoscan®, marketed and used among diabetic patients or not for the detection of violations neuropathic (cf. references and CE certificate attached to the dossier).

The Thermotest® is also marketed and used in diabetic and non-diabetic patients (see references and CE certificate attached to the dossier).

Our center has gained experience of these techniques for the detection of peripheral neuropathy in several patient populations (diabetes and cancer in particular); manipulators (doctors and technicians) are trained in these techniques.

Data collection for each patient:

* Clinical data:

  * Age
  * Gender
  * BMI
  * Size
  * Weight
  * Waist
  * Hips
  * Report on waist hips
  * Blood pressure: systolic, diastolic, mean
  * Score Questionnaire DN4 (presence or absence of neuropathic pain)
  * Score Uens
* electrophysiological data

  o skin conductance (μSiemens) measured by the Sudoscan®
* Plants Average feet (right, left)

  * Thermotest®: average score of sensitivity threshold to pain in plantar warm level (average of the soles of both feet).
  * Electromyography:
* Sensitive Conduction:

  • sural nerve left and right (lateral malleolus collection, antidromic calf stimulation), radial nerve left and right (wrist collection, antidromic stimulation forearm)
  * Amplitude (mV)
  * VCS (sensory conduction velocity m / s)
* Motor Conduction:

  * Sciatic nerve popliteal internal right and left (short collection flexor hallucis longus, ankle stimulation)

    * distal motor latency (ms)
    * amplitude of CMAP (mV)
    * Latency wave F shortest (ms).
  * tibial nerve left and right anterior (short collection extensor hallucis longus, ankle stimulation under neck of the fibula, above-neck of the fibula)

    * distal motor latency (ms)
    * Amplitude of PGAM 3 to stimulation points (mV)
    * PNT leg and neck of the fibula (m / s).
    * Latency wave F shortest (ms).
* EMG needle:

  * Muscles studied: tibialis anterior right, wide left inner, right brachioradialis.
  * Rest Activities: yes / no
  * Activation Pattern:

    * normal Interferential
    * Intermediate with poor temporal summation
    * Poor with temporal summation
    * Single with temporal summation
* Biological data:

  * Fasting glucose
  * HbA1c
  * Triglycerides
  * Total cholesterol
  * HDL cholesterol
  * LDL Cholesterol
  * uricaemia
  * SGOT, SGPT, gammaGT
  * urea, creatinine
  * creatinine clearance
  * Microalbuminuria on sample
  * serum folate,
  * vitamins D, B1 and B12,
  * calcemia
  * albumin
  * NFS, CRP
  * Electrophoresis + plasma protein immunofixation.

Data processing :

For each subject will be awarded an identifier (original name and surname - year of birth) and the data will be entered on a computer file which will be sent to the statistician in charge of analyzing the GHPSJ site. There will be no exchange of personal data.

Statistical analysis :

The patient will be considered to have a small fiber neuropathy, symptomatic or not, when the skin conductance of chloride ions will be below the threshold for 60μSiemens soles. The prevalence shall be calculated from that definition.

Stratified by age will be made during the statistical analysis.

A test will be performed to analyze the statistical relationship between:

Skin conductance AND

* BMI,
* size,
* Girth
* Waist circumference ratio / hip circumference
* Sex,
* DN4 score,
* The score Uens,
* The biological parameters studied: fasting blood glucose, HbA1c, total cholesterol, HDL cholesterol, triglycerides, CRP, serum uric acid.
* Threshold of pain sensitivity warm on the feet by Thermotest.
* Type of surgery for surgical patients.

Ethics / Regulatory:

The patient will be informed orally of the objective of the study, a leaflet it will also be provided (attached); its information and not be drawn opposition in his file.

All tests are part of the normal patient care. The ethics of the CPP Ile de France approved this study on march 15th 2015. The manager research center will be the hospital group Paris Saint-Joseph (GHPSJ).

partnerships

Impeto the company, the manufacturer will provide Sudoscan® (loan agreement) the machine for the duration of the study.

GHPSJ ensure the neurologist time, diabetologist, biologist and ARC necessary and will provide the Thermotest® machine for the duration of the study.

Conflicts of interest :

No conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patients:
* BMI 35-55 kg / m²
* Male or female
* Age> 18 and <60 years
* Consultant for the first time at the Centre of obesity of Paris Saint Joseph Hospital Group.

Exclusion Criteria:

* Diabetes known treaty
* Co-morbidity related to obesity: heart disease, respiratory failure
* Other causes of peripheral neuropathy:
* Alcohol Poisoning
* Renal failure (clearance ≤ 60 mL / min)
* Infection HIV, hepatitis B, C
* Deficiencies vitamins B1, B6, B12, folate
* Treatment with vitamin B6
* thyroid disease antecedent
* Previous history of autoimmune disease
* Previous history of cancer
* Previous history of neurotoxic treatment (chemotherapy, etc. see list provided in annex)
* ICU hospitalization antecedent> 48 hours.
* known history of peripheral neuropathy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Chlorine ion production change | at inclusion then 1 month, 3 months, 6months and 12 months after surgery
  Patients will be a measure of impedance of the skin to products chlorine ions by the sweat glands via the Sudoscan® Device, marketed and used among diabetic patients or not for the detection of violations neuropathic (cf. references and CE certificate attached to the dossier)
Assessment of Temperature changing sensitivity | At inclusion then 1 month, 3 months, 6months and 12 months after surgery
  Patients will be measured their sensitivity to temperature changing using the Thermotest Device

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu ZUBER, MD, Principal Investigator — Groupe Hospitalier Paris Saint-Joseph (FRANCE)
Locations (1):
- Groupe Hopitalier Paris Saint Joseph Service de neurologie, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Smith AG, Lessard M, Reyna S, Doudova M, Singleton JR. The diagnostic utility of Sudoscan for distal symmetric peripheral neuropathy. J Diabetes Complications. 2014 Jul-Aug;28(4):511-6. doi: 10.1016/j.jdiacomp.2014.02.013. Epub 2014 Mar 6. PMID 24661818
- [Result] Kopelman PG. Obesity as a medical problem. Nature. 2000 Apr 6;404(6778):635-43. doi: 10.1038/35007508. PMID 10766250
- [Result] Herman RM, Brower JB, Stoddard DG, Casano AR, Targovnik JH, Herman JH, Tearse P. Prevalence of somatic small fiber neuropathy in obesity. Int J Obes (Lond). 2007 Feb;31(2):226-35. doi: 10.1038/sj.ijo.0803418. Epub 2006 Jun 13. PMID 16770330
- [Result] Philippi N, Vinzio S, Collongues N, Vix M, Boehm N, Tranchant C, Echaniz-Laguna A. [Peripheral neuropathies after bariatric surgery]. Rev Neurol (Paris). 2011 Aug-Sep;167(8-9):607-14. doi: 10.1016/j.neurol.2011.01.011. Epub 2011 Apr 22. French. PMID 21514611
- [Result] Thaisetthawatkul P, Collazo-Clavell ML, Sarr MG, Norell JE, Dyck PJ. A controlled study of peripheral neuropathy after bariatric surgery. Neurology. 2004 Oct 26;63(8):1462-70. doi: 10.1212/01.wnl.0000142038.43946.06. PMID 15505166
- [Result] Sumner CJ, Sheth S, Griffin JW, Cornblath DR, Polydefkis M. The spectrum of neuropathy in diabetes and impaired glucose tolerance. Neurology. 2003 Jan 14;60(1):108-11. doi: 10.1212/wnl.60.1.108. PMID 12525727
- [Result] Devigili G, Tugnoli V, Penza P, Camozzi F, Lombardi R, Melli G, Broglio L, Granieri E, Lauria G. The diagnostic criteria for small fibre neuropathy: from symptoms to neuropathology. Brain. 2008 Jul;131(Pt 7):1912-25. doi: 10.1093/brain/awn093. Epub 2008 Jun 4. PMID 18524793
- [Result] Casellini CM, Parson HK, Richardson MS, Nevoret ML, Vinik AI. Sudoscan, a noninvasive tool for detecting diabetic small fiber neuropathy and autonomic dysfunction. Diabetes Technol Ther. 2013 Nov;15(11):948-53. doi: 10.1089/dia.2013.0129. Epub 2013 Jul 27. PMID 23889506